CLINICAL TRIAL: NCT04560777
Title: Exploring the Use of the Cognitive Orientation to Daily Occupational Performance Approach (CO-OP) With Children, Teenagers and Young Adults With Executive Functions Deficits Following Severe Acquired Brain Injury
Acronym: REFECO-OP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopitaux de Saint-Maurice (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Hôpital Civil de Strasbourg (Unknown); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHRIP-19-0074
Record Dates: First submitted 2020-09-15; First posted 2020-09-23 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Acquired Brain Injury
Keywords: Cognitive Orientation to daily Occupational Performance; rehabilitation; executive functions; child acquired brain injury; teenagers; young adults; acquired brain injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: Single case experimental study design with multiple baselines across individuals and behaviors.
  Randomization:
  1. Which patient starts when the COOP sessions?
  2. What are the possible starting points for the 3 goals to be worked on?
  3. Which of the 4 goals ABCD is assigned to which goal number? The most important goal (A) will necessarily be worked on first. We will draw lots to determine the order in which the goals will be worked on and which goal will be designated as the control goal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): CO-OP intervention
  Interventions: Other: CO-OP intervention

INTERVENTIONS:
Other: CO-OP intervention — The general structure of the intervention will follow the original key principles of CO-OP, with some adjustments to adapt it to the specificities of the ABI population (14 CO-OP sessions vs 10 in the original protocol).
  The global strategy will be taught to the participant at the first session. The following sessions will be consisted of an process of implementation of the global strategy in the context of guided discovery to identify domain specific strategies to overcome performance ''breakdowns" the participant will be experiencing when performing the self-selected tasks. In addition, "homework" will be assigned to encourage the application and practice of the cognitive strategies discovered during the intervention sessions. Parents will be invited to attend the sessions if it will be possible for them. In any case, the global strategy, as well as the progress of the child, will be explained to the parents.

SUMMARY:
Acquired brain injury (ABI) in childhood are the cause of disabling motor, cognitive and behavioural disorders, with severe consequences on the later development of autonomy and learning, with long-term repercussions on independence for activities of daily living, and social and professional integration.

Among cognitive disorders, executive function (EF) deficits are among the most frequent and disabling, with major consequences on the development of autonomy and the course of schooling and learning.

The Cognitive Orientation to daily Occupational Performance (CO-OP) could be an interesting approach for the rehabilitation of these consequences. CO-OP is a performance-based treatment approach for children and adults who experience difficulties performing the skills they want to, need to or are expected to perform. CO-OP is a specifically tailored, active client-centered approach that engages the individual at the meta-cognitive level to solve performance problems. Focused on enabling success, the CO-OP approach employs collaborative goal setting, dynamic performance analysis, cognitive strategy use, guided discovery, and enabling principles.

It has been shown to be effective in a variety of populations, but has been little explored in children with ABI. The hypothesis that CO-OP is effective in improving the occupational performance and executive functioning of these children on a daily basis is emerging, but needs to be confirmed. This study falls within this framework.

Primary objective:

1. To measure the distance maintenance of the knowledge acquired through rehabilitation, as well as the generalization and transfer into everyday life.

   1. Maintenance of acquired knowledge
   2. Generalization and transfer
   3. Impact of a consolidation session on generalization and transfer

   Secondary objectives:
2. Gather the experience of family members/caregivers in accompanying their child in the CO-OP process outside of rehabilitation sessions.
3. Establish the parental educational style and identify whether there is a link between the parental educational style and the commitment of the family members/caregivers.

DETAILED DESCRIPTION:
Twelve participants will be included (aged 8 to 21 years old). Participants will have different assessment times, before, during and after the CO-OP intervention (immediate post-intervention, 2, 4 and 6-months post-intervention). Parents will be asked to answer questionnaires and interview and to participate in certain CO-OP sessions, if they can.

They will choose four objectives (problematic everyday life activities they want to improve). Three will be worked on in CO-OP sessions, the fourth will be the control objective.

The duration of the baseline, as well as the order of introduction of the objectives and the starting point of the objectives, are randomized.

Participants will have 14 sessions of rehabilitation with the CO-OP approach (2 sessions per week for 7 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Child/adolescent/young adult aged between 8 and 21 years old, hospitalized in the Acquired Neurological Pathologies Service of the Saint-Maurice Hospitals or in the Medical and Pedagogical Centre for Adolescents of Neufmoutiers-en-Brie, and possibly schooled in this service.
2. Diagnosis of acquired brain injury, for at least 6 months.
3. Child/adolescent/young adult presenting executive function deficits as determined by the neuropsychological assessment (standardized tests and/or questionnaire).
4. Vision and hearing normal or sufficient to communicate effectively (with appropriate correction if necessary).
5. Having sufficient speaking and comprehension skills to communicate effectively and accurately.
6. Enrollment in a Medicare plan or eligible beneficiary.
7. Agreement of the child/young person and informed consent expressed by the holders of parental authority. Consent of the young adult (18-21 years of age).

Exclusion Criteria:

1. Non-Francophone child/teenager/young adult and/or non-Francophone parents.
2. With an intellectual disability (total IQ <70), or severe impairment in comprehension, memory or attention, not compatible with understanding the goals of the rehabilitation and participation in 45-minute sessions.
3. Neurological, psychiatric, genetic or learning disorder diagnosed prior to the occurrence of the acquired brain injury.
4. Severe anxiety and/or depressive disorder diagnosed that is not compatible with participation in the study.
5. Inability to commit until the end of the CO-OP rehabilitation phase (e.g., planned relocation, planned hospital discharge before the end of the 14 CO-OP sessions, i.e., 10 weeks including baseline and CO-OP rehabilitation).
6. Major subject under guardianship or curatorship.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Assessment of Goal Attainment Scaling (GAS) change | Baseline to 6-months post-intervention (Two times per week during baseline and intervention phase for each 4 chosen-goal ; one time at 2, 4 and 6-months post-intervention)
  Goal Attainment Scaling (GAS) is a method for writing personalized evaluation scales in order to quantify progress toward defined goals.
  GAS methodology consists in:
  * Defining a rehabilitation goal;
  * Choosing an observable behaviour that reflects the degree of goal attainment;
  * Defining the patient's initial level with respect to the goal;
  * Defining five goal attainment levels (ranging from a ''no change'' to a ''much better than expected outcome'');
  * Evaluating the patient after a defined time interval;
  * Calculating the overall attainment score for all the rehabilitation goals. A five-point scale is used: ''-2'' is the initial pretreatment (baseline) level, ''-1'' represents progression towards the goal without goal attainment, ''0'' is the expected level after treatment, (and therefore, the ''most likely'' level after treatment), ''+1'' represents a better outcome than expected, and ''+2'' is the best possible outcome that could have been expected for this goal.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Before baseline, at immediate post-intervention, at 2, 4 and 6-months post-intervention.
  This semi-structured interview helps children/parents identify problematic occupations in different daily areas. COPM will be used: (1) To determine (only with the child) the 4 problematic occupations identified as the most important (3 will be used as target goals, while the 4 will serve as a control goal); (2) To determine changes in occupational performance in self-selected goals: children and parents will rated their performance and satisfaction associated with these 4 occupations.
  Performance and satisfaction are rated by children and parents on a scale of 1 to 10 (1= not at all able to perform the activity (performance) / not at all satisfied with the way the activity is performed (satisfaction); 10 = perfectly able to perform the activity (performance) / perfectly satisfied with the way the activity is performed (satisfaction). A difference of 2 points between pre- and post-intervention is clinically significant.
Behavior Rating Inventory of Executive Function (BRIEF) | Minimum 3-maximum 6 assessments during the baseline (according the duration of the baseline), week 2, 4 and 6 during the intervention, at immediate post-intervention, at 2, 4 and 6-months post-intervention.
  The parent and teacher report forms of the Behavior Rating Inventory of Executive Function (BRIEF, or BRIEF-A for adults'version) provide an ecological assessment of executive functioning through its repercussions in family and school context. Currently, this questionnaire is the best validated and most widely used in children in various congenital, developmental or acquired conditions.
  The outcome measure is the Global Executive Composite score (GEC) T-Scores (Mean: 50; SD: 10; clinical range cutoff: T-Scores≥65).
Évaluation des Pratiques Éducatives Parentales (EPEP, Parental Childrearing Behavior Scale for French-Speaking Parents, Children, and Adolescents) | one time before baseline
  The EPEP represents an efficient solution to the search for conceptually and psychometrically sound instruments to assess parents' child-rearing behavior. A 5-point Likert-type scale is provided for each item ranging from "never" "to always" (explaining to parents that there are no right or wrong answers). The results are obtained by averaging the scores per subscale (8 subscales). The purpose of this evaluation is to define the parenting educational style: there are not a better or worse outcome per se.
Questionnaire Engagement des Proches | week 2, 4 and 6 during the intervention
  The objective of this questionnaire is to collect information on the use of CO-OP by family caregivers with the participant, outside of rehabilitation sessions. No scale of score, just a collection of factual facts.
Entretien Engagement des Proches | immediate post-intervention, 4 and 6 months-post-intervention
  The objective of this interview is to collect information on the experience of use of CO-OP by family caregivers with the participant, outside of rehabilitation sessions. No scale of score, the interviews will be analyzed according to a qualitative description.

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde CHEVIGNARD, PhD, Study Director — Hopitaux de Saint-Maurice
Locations (2):
- France (2):
  - Centre Médical et Pédagogique pour Adolescents, Neufmoutiers-en-Brie
  - Hôpitaux de Saint-Maurice, Saint-Maurice

IPD SHARING:
Plan to Share IPD: Undecided
We think it would be interesting to share the IPD with other researchers (especially Canadian researchers), but we have not yet defined the terms of this sharing.

REFERENCES:
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Krasny-Pacini A, Hiebel J, Pauly F, Godon S, Chevignard M. Goal attainment scaling in rehabilitation: a literature-based update. Ann Phys Rehabil Med. 2013 Apr;56(3):212-30. doi: 10.1016/j.rehab.2013.02.002. Epub 2013 Feb 28. PMID 23562111
- [Background] Scammell EM, Bates SV, Houldin A, Polatajko HJ. The Cognitive Orientation to daily Occupational Performance (CO-OP): A scoping review. Can J Occup Ther. 2016 Oct;83(4):216-225. doi: 10.1177/0008417416651277. Epub 2016 Jun 14. PMID 27301479
- [Derived] Manolov R, Lebrault H, Krasny-Pacini A. How to assess and take into account trend in single-case experimental design data. Neuropsychol Rehabil. 2024 Apr;34(3):388-429. doi: 10.1080/09602011.2023.2190129. Epub 2023 Mar 24. PMID 36961228